CLINICAL TRIAL: NCT03843190
Title: Changes in Weight and Physical Function for Older African American Women in a National, Nonprofit, Community-Based, Peer-Led, Weight Loss Program
Brief Title: Healthy Me: A Program for Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100588; R01AG058725 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: weight loss; african american women; physical function
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take Off Pounds Sensibly (TOPS) (Experimental): This group will receive TOPS intervention at the start of the study.
  Interventions: Behavioral: Take of Pounds Sensibly (TOPS)
- Waitlist control (Other): This group will be the control group for 6 months. Then at the completion of the study they will receive the vouchers to participate in TOPS chapters in the community.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Take of Pounds Sensibly (TOPS) — Dietician-facilitated classes
  Arms: Take Off Pounds Sensibly (TOPS)
Other: Waitlist Control — At end of study, offered peer-led classes to attend.
  Arms: Waitlist control

SUMMARY:
The first phase of the study is a feasibility survey of eligible participants, completed prior to initiating the intervention. The intervention consists of a 6-month 1:1 randomized trial with a waitlist control that recruits 120 older AA women. The rationale for these aims is that the successful completion is expected to provide evidence that a community-based, peer-led weight loss program with a national infrastructure can help a vulnerable, underserved population lose weight and improve their physical function. For older, obese, frail individuals, this could improve their CVD risk factors, quality of life, enhance their health; reduce their healthcare utilization, illness, and disability; and decrease their adverse geriatric outcomes. After completing these aims, the investigators expect that they will have proven that the community-based, peer-led weight loss program can improve both weight and physical function among older, obese AA women. This also could help other demographic groups with obesity and poor physical function. Eventually, it could help older adults maintain their health and independence in the community

DETAILED DESCRIPTION:
Older African American (AA) women have the highest prevalence of both obesity and frailty. In academic, expert-led interventions, obese, frail, older individuals both lost weight and improved their physical function. However, because of high personnel costs and nonexistent nationwide infrastructure, large-scale implementation of these interventions is impractical. The long-term goals are to eliminate the health disparities of obesity and frailty in older AA women. This proposal's overall objective is to determine the effects of a low-cost, community-based, peer-led weight loss program with a national infrastructure on obesity, physical function, and healthcare utilization in older AA women. To treat obesity and frailty in older AA women, it is critical to test a weight loss intervention that 1) has preliminary evidence of benefit; 2) is acceptable to older AA women; 3) is affordable; and 4) can be broadly disseminated. Take Off Pounds Sensibly (TOPS) is a national, nonprofit, community-based, peer-led weight loss program that meets these criteria. First, the applicant's retrospective database analyses of TOPS showed two important results: 1) Participants who renew their annual membership lose and maintain significant weight loss (SWL) for up to 7 years; and 2) Compared to their younger counterparts, older women are more likely to achieve SWL. Second, the applicant started three TOPS chapters for older AA women in a successful pilot study. Though the study ended in 2012, one of the chapters is still active almost 6 years later. Third, TOPS is affordable; it only costs $120 annually. Finally, TOPS has a nationwide infrastructure with chapters in all 50 states. Since obese, frail, older individuals in academic, expert-led weight loss interventions can improve their physical function, the central hypothesis is that a low cost, community-based, peer-led weight loss program with a national infrastructure can provide SWL, improved physical function, and lower healthcare utilization for AA women, an underserved, vulnerable population. The rationale for the proposed research is that TOPS and academic, expert-led weight loss interventions share components critical to successful weight loss; therefore, TOPS can deliver similar outcomes. The central hypothesis will be tested by pursuing the following aims in obese, frail, older AA women: Determine the effect of TOPS on 1) weight change and cardiovascular disease risk factors; 2) physical function and quality of life; and 3) healthcare utilization. This project is innovative because it uses a "community to academia" approach to treat the health disparities; our study population focuses on older AA women with decreased physical function; our outcomes focus on weight, physical function, and healthcare utilization; and our unique study settings. The proposed research is significant because determining the real-world effectiveness of the TOPS program and its impact on weight, physical function, and healthcare utilization in AA women can have a widespread impact on the older population at large. Thus, it has the potential to reduce adverse geriatric outcomes among all older individuals.

ELIGIBILITY:
Inclusion Criteria:

* African American women aged ≥55
* BMI ≥27 kg/m2
* Stable body weight (± 2 kg for 6 months prior to study)
* Sedentary (not exercising more than 1 hour per week)
* Must have a primary care provider and provide contact information

Conditional Inclusion Criteria:

Participants with type 2 diabetes on insulin or sulfonylureas will be allowed to participate in the study only if their providers agree to manage the changing medications requirements associated with possible weight loss by signing a "Permission to Participate" form. It is important to include patients with type 2 diabetes on insulin and sulfonylureas because these participants can benefit greatly from weight loss.

Exclusion Criteria:

* Type 2 diabetes on insulin or sulfonylureas without provider approval
* current cancer diagnosis
* Provider did not approve participation
* use of medications thought to effect metabolism, body weight, energy expenditure, or appetite
* major psychiatric disorder
* current moderate to severe symptoms of depression
* dementia
* neurological conditions causing functional limitations
* unstable medical illness such as unstable angina, recent MI, or congestive heart failure class III-IV
* terminal medical conditions
* Currently enrolled in a weight loss program

Ages: 55 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — African-American women
Enrollment: 119 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Weight change | up to 6 months
  Percent of weight loss over 6 months

SECONDARY OUTCOMES:
Cardiovascular Disease (CVD) risk factors as measured by Blood pressure (BP) | up to 6 months
Cardiovascular Disease (CVD) risk factors as measured by Waist circumference (WC) | up to 6 months
Cardiovascular Disease (CVD) risk factors as measured by Hemoglobin A1c (HA1c) | up to 6 months
Cardiovascular Disease (CVD) risk factors as measured by Lipids | up to 6 months
Quality of Life (QoL) as measured by 36-item short form survey (SF-36) | up to 6 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Healthcare Utilization as measured by surveys of inpatient stays and outpatient visits | up to 6 months
Physical Function as measured by Short physical performance battery (SPPB) | up to 6 months
  The Short Physical Performance Battery (SPPB) is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults. Scores range from zero to 12 possible points. Lower score are associated with lower function.
Physical Function as measured by 8-ft up and go | up to 6 months
  The 8-foot up-and-go test is a timed test that measures balance, agility, and speed while walking or moving. Higher times are associated with worse physical function.
Physical Function as measured by Isometric hand grip | up to 6 months
  Decreased grip strength is a predictor of adverse outcomes in older adults.
Physical Function as measured by 30-second chair stands | up to 6 months
  Counts the number of time a participants goes from sitting to standing in 30 seconds. Tests leg strength and endurance. Higher number associated with higher leg strength and endurance.
Physical Function as measured by 6-minute walk test | up to 6 months
  Measures distance walked in 6 minutes and assesses aerobic capacity and endurance. higher number indicate higher aerobic capacity and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Nia S Mitchell, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT03843190/ICF_000.pdf